CLINICAL TRIAL: NCT05611385
Title: High Incidence of Adult Respiratory Distress Syndrome Associated With Amphetamine Use in the Burn Population
Brief Title: Amphetamine Induced Adult Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-24
Record Dates: First submitted 2022-10-26; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Burns; Acute Lung Injury; Acute Respiratory Distress Syndrome; Methamphetamine Abuse
MeSH Terms: conditions — Burns; Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive for Amphetamine: Patients admitted to the burn unit that are positive for amphetamine
  Interventions: Other: Difference in development of Acute Lung Injury in Amphetamine positive and negative patients
- Negative for Amphetamine: Patients admitted to the burn unit that are negative for amphetamine
  Interventions: Other: Difference in development of Acute Lung Injury in Amphetamine positive and negative patients

INTERVENTIONS:
Other: Difference in development of Acute Lung Injury in Amphetamine positive and negative patients — No Intervention

SUMMARY:
Methamphetamine and amphetamine has various cardiovascular and central nervous system effects. Long-term use is associated with many adverse health effects including cardiomyopathy, hemorrhagic, and ischemic stroke. Death is usually caused by cardiovascular collapse and while amphetamine abuse has been considered as a potential cause of acute respiratory distress syndrome, the reports are usually anecdotal. This investigation considers reviewing individuals with few to zero medical conditions who develop acute respiratory distress syndrome and are methamphetamine positive

DETAILED DESCRIPTION:
Methamphetamine and amphetamine has various cardiovascular and central nervous system effects. Initially prescribed in the 1930s for respiratory ailments such as asthma, current clinical indications of amphetamine range from treatment of attention deficit hyperactivity disorder to narcolepsy. The mechanism of action is primarily potentiation of release of monoamine neurotransmitters, mainly dopamine and norepinephrine, from presynaptic nerve endings into the synaptic space, in addition to attenuation of monoamine metabolism by inhibiting monoamine oxidase. This in turn leads to an increase in sympathetic tone by alpha and beta adrenergic receptor activation, resulting in elevations in heart rate, respiratory rate, and vascular tone. Long-term use is associated with many adverse health effects including cardiomyopathy, hemorrhagic and ischemic stroke. Other long-term associations include increased violent behavior, documented increased motor vehicle accidents, and clandestine manufacturing of the drug.

Methamphetamine has also been associated with deleterious effects on society as a whole; it is credited as a cause of increase in rates of crime, abuse, and unemployment, and associated with great economic burden. A significant portion of healthcare resources consumed are rooted in the emergency department, particularly in trauma. Studies previously performed have demonstrated that methamphetamine use among patients that present to trauma centers has been continually increasing. Death is usually caused by cardiovascular collapse and while amphetamine abuse has been considered as a potential cause of acute respiratory distress syndrome, the reports are usually anecdotal. This investigation considers reviewing individuals with few to zero medical conditions who develop acute respiratory distress syndrome and are methamphetamine positive

ELIGIBILITY:
Inclusion Criteria:

* Total body surface area burns between 20% and 60% admitted to the burn unit

Exclusion Criteria:

* Under 18 years of age
* Burns outside of the inclusion ratio

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was completed at Arrowhead Regional Medical Center County Burn Center in Colton, California, which operates as the only burn center for San Bernardino, Inyo, Mono and Riverside Counties. ARMC covers one of the largest geographical areas in the United States. Due to the high prevalence of methamphetamine use, this location sees a high incidence of burn patients who either use amphetamine or are the result of methamphetamine lab explosions.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Inhalation Injury | 24 hours
  Documentation on admission of inhalation injury as defined by burned nasal hairs, burned facial skin, and carbonaceous sputum after admission to the hospital within the first 24 hours.
Total Burn Surface Area | 24 hours
  The total burn surface area of the patient on arrival to the hospital assessed within the first 24 hours. With respect to the total burn surface area recorded only 2nd degree burns will be considered as defined as burns that affect the epidermis and dermis.
Length of hospital stay | 180 days
  The total length of hospitalization of individuals with burns and acute respiratory distress syndrome with a max of 180 days from admission.
Stroke Volume | Collected in the first 5 days after admission
  Measurement of cardiovascular parameter (stroke volume) of patients with acute respiratory distress syndrome and total burn surface area between 20%-60% in the first 5 days of admission to the hospital.
Cardiac Output | Collected in the first 5 days after admission
  Measurement of cardiovascular parameter (cardiac output) of patients with acute respiratory distress syndrome and total burn surface area between 20%-60% in the first 5 days of admission to the hospital.
Central Venous Pressure | Collected in the first 5 days after admission
  Measurement of cardiovascular parameter (central venous pressure) of patients with acute respiratory distress syndrome and total burn surface area between 20%-60% in the first 5 days of admission to the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Aldin Malkoc, MD, Study Chair — Arrowhead Regional Medical Center; David T Wong, MD, Principal Investigator — Arrowhead Regional Medical Center
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Busto U, Bendayan R, Sellers EM. Clinical pharmacokinetics of non-opiate abused drugs. Clin Pharmacokinet. 1989 Jan;16(1):1-26. doi: 10.2165/00003088-198916010-00001. PMID 2565176
- [Background] Gonzales R, Mooney L, Rawson RA. The methamphetamine problem in the United States. Annu Rev Public Health. 2010;31:385-98. doi: 10.1146/annurev.publhealth.012809.103600. PMID 20070191
- [Background] Neeki MM, Kulczycki M, Toy J, Dong F, Lee C, Borger R, Adigopula S. Frequency of Methamphetamine Use as a Major Contributor Toward the Severity of Cardiomyopathy in Adults </=50 Years. Am J Cardiol. 2016 Aug 15;118(4):585-9. doi: 10.1016/j.amjcard.2016.05.057. Epub 2016 May 29. PMID 27374605
- [Background] Kaye S, McKetin R, Duflou J, Darke S. Methamphetamine and cardiovascular pathology: a review of the evidence. Addiction. 2007 Aug;102(8):1204-11. doi: 10.1111/j.1360-0443.2007.01874.x. Epub 2007 Jun 12. PMID 17565561
- [Background] Jafari Giv M. Exposure to Amphetamines Leads to Development of Amphetamine Type Stimulants Associated Cardiomyopathy (ATSAC). Cardiovasc Toxicol. 2017 Jan;17(1):13-24. doi: 10.1007/s12012-016-9385-8. PMID 27663745
- [Background] Weir EK, Reeve HL, Huang JM, Michelakis E, Nelson DP, Hampl V, Archer SL. Anorexic agents aminorex, fenfluramine, and dexfenfluramine inhibit potassium current in rat pulmonary vascular smooth muscle and cause pulmonary vasoconstriction. Circulation. 1996 Nov 1;94(9):2216-20. doi: 10.1161/01.cir.94.9.2216. PMID 8901674